CLINICAL TRIAL: NCT05943522
Title: A Post Approval Surveillance of Scemblix® (Asciminib) in Patients With Chronic Myeloid Leukemia (CML) in Korea
Brief Title: Asciminib RMP Study
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001A2006
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Scemblix; Asciminib; CML; Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — asciminib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Asciminib: Patients prescribed with Asciminib at physicians' discretion as per locally approved label under usual clinical practice
  Interventions: Other: Asciminib

INTERVENTIONS:
Other: Asciminib — There is no treatment allocation. Asciminib will be prescribed by the physician as per locally approved label. No drug will be dispensed from Novartis
  Other Names: Scemblix

SUMMARY:
This study is a prospective, open-label, multi-center, non-comparative, observational study to assess safety and effectiveness of Asciminib in the real-world clinical setting in Korean Chronic myeloid leukemia (CML) patients.

DETAILED DESCRIPTION:
The dosage and duration of treatment may be considered and decided by the investigator in accordance with prescribing information of Asciminib.

This study will enroll all patients by total enumeration for those prescribed with Asciminib at physicians' discretion as per locally approved label under usual clinical practice for 2 years after the market launch.

ELIGIBILITY:
Inclusion criteria

1. Adult patients diagnosed with Ph+ CP-CML and currently receiving or going to receive Scemblix® treatment according to locally approval label
2. Patients who are willing to provide written informed consent prior to study enrollment

Exclusion criteria

1. Patients with contraindication according to locally approved label of Scemblix®
2. Patients who receive or are going to receive any investigational medicine during the observation period

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are going to receive Scemblix® for the first time or those who are currently taking Scemblix® per clinical judgment are eligible and will be prescribed with Scemblix® under routine medical practice.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with an AE / ADR | 24 weeks
  Percentage of participants with an adverse event (AE)/ adverse drug reaction (ADR)
Percentage of participants with a SAE / SADR | 24 weeks
  Percentage of participants with a serious AE (SAE)/ serious ADR (SADR)
Percentage of participants with an UAE/ UADR | 24 weeks
  Percentage of participants with an unexpected AE (UAE)/ unexpected ADR (UADR)
Percentage of participants with a SUAE/ SUADR | 24 weeks
  Percentage of participants with a serious unexpected AE (SUAE)/ serious unexpected ADR (SUADR)

SECONDARY OUTCOMES:
Major molecular response rate | week 12, week 24
  Major molecular response (MMR) rate at week 12 and week 24
Molecular response 4 rate | week 12, week 24
  Molecular response 4 (MR4) rate. Molecular response (MR) is a Breakpoint Cluster Region protein Tyrosine-protein kinase ABL1 (BCR-ABL1) transcript that is assessed by real-time quantitative PCR (RQ-PCR) in the blood at screening. Molecular response levels are indicated with a superscript indicating the log reduction from the standardized baseline, corresponding to 100% on the international scale (IS).
Molecular response 4.5 rate | week 12 ,week 24
  Molecular response 4.5 (MR4.5) rate. Molecular response (MR) is a Breakpoint Cluster Region protein Tyrosine-protein kinase ABL1 (BCR-ABL1) transcript that is assessed by real-time quantitative PCR (RQ-PCR) in the blood at screening. Molecular response levels are indicated with a superscript indicating the log reduction from the standardized baseline, corresponding to 100% on the international scale (IS).
Number of participants with CCyR and/or BCR-ABL1 IS<1% | week 12,week 24
  Complete cytogenetic response (CCyR) rate and/or BCR-ABL1 IS<1%.
  A complete cytogenetic response (CCyR) is defined as absence of the Ph (0%) among at least 20 cells in metaphase in a bone marrow aspirate.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- South Korea (9):
  - Novartis Investigative Site, Wŏnju, Gangwon-do
  - Novartis Investigative Site, Uijeongbu-si, Gyeonggi-do
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Jeollanam
  - Novartis Investigative Site, Pusan
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu

IPD SHARING:
Plan to Share IPD: No